CLINICAL TRIAL: NCT06947252
Title: Validation of Food Allergies in Pediatric Atopic Dermatitis Patients Practicing Food Avoidance
Brief Title: Frequency of Food Allergy Confirm by Oral Food Challenge Among Foods Avoidance in Atopic Dermatitis Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 998/2567(IRB3)
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Food Allergies
Keywords: Atopic dermatitis; Food allergies; Oral food challenge test
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atopic dermatitis children that avoid some foods (Experimental): Oral food challenge test
  Interventions: Diagnostic Test: Oral food challenge test

INTERVENTIONS:
Diagnostic Test: Oral food challenge test — Oral food challenge test at home or in the hospital

SUMMARY:
Atopic dermatitis can be caused by several factors, including food allergy. Currently, the diagnosis of food allergy often performing skin tests and measuring specific IgE foods that many studies have shown that about 53% of children with atopic dermatitis have food sensitization, result in avoidance of food intake. But only 15% are confirmed to have a true food allergy, so the purpose of our study is to find the prevalence of food allergy in Thai children with atopic dermatitis who are avoiding some foods, using the oral food challenge to confirm the diagnosis to reduce unnecessary food avoidance and prevent complications from inappropriate dietary restrictions

DETAILED DESCRIPTION:
All subject in this study were patients with history of atopic dermatitis and avoid at least 1 food of egg yolk, egg white, cow milk, peanut, wheat or soy. All of them will undergo a blood testing for specific IgE foods to assess whether they can resume consuming that particular food or they must perform oral food challenge test in hospital to evaluate whether they truly have a food allergy or should continue to avoid that food.

The primary outcome was to study frequency of food allergy confirm by oral food challenge among foods avoidance in atopic dermatitis children, focusing on the 6 major food allergens in the Thai children: egg yolk, egg white, cow milk, peanut, wheat and soy. Other outcomes were study type of food reaction after oral food challenge test in atopic dermatitis children (IgE mediated, delayed type: AD flare)

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 6 years
* Age ≤ 6 years with diagnosis of atopic dermatitis c
* Now parent report them avoid at least 1 food of egg yolk, egg white, cow milk, peanut, wheat or soy

Exclusion Criteria:

* Specific IgE food > 95%PPV (73-74%PPV in wheat, soy)
* Patients with uncontrolled asthma/ atopic dermatitis
* Patients who had been treated with some other immunotherapy e.g. SCIT, OIT
* Patients with delayed developmental problem or mental disorder
* Patient use beta-blocker, ACEI, ARB
* Patient who unable to follow up

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of food allergy among foods avoidance in atopic dermatitis children | 7 days
  Frequency of food allergy confirm by oral food challenge among foods avoidance in atopic dermatitis children, focusing on the 6 major food allergens in the Thai children: egg yolk, egg white, cow milk, peanut, wheat, soy

SECONDARY OUTCOMES:
Type of food reaction after oral food challenge test in atopic dermatitis children | 7 days
  Type of food reaction after oral food challenge test in atopic dermatitis children divide to IgE mediated or delayed type (AD flare)

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, Principal Investigator — Mahidol University, Siriraj Hospital, Thailand
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eapen AA, Kloepfer KM, Leickly FE, Slaven JE, Vitalpur G. Oral food challenge failures among foods restricted because of atopic dermatitis. Ann Allergy Asthma Immunol. 2019 Feb;122(2):193-197. doi: 10.1016/j.anai.2018.10.012. Epub 2018 Oct 14. PMID 30326323